CLINICAL TRIAL: NCT03672981
Title: Pilot Study of a Resistance Training Intervention in Adolescent and Young Adult Hematopoietic Cell Transplant Survivors
Brief Title: Resistance Training Program and Cardiovascular Exercise in Increasing Muscle Mass in Adolescent and Young Adult Stem Cell Transplant Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Conquer Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10046; NCI-2018-01254 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10046 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1001740 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-07-19; First posted 2018-09-17 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (aerobic exercise and resistance training) (Experimental): Patients undergo moderately intense aerobic/cardiovascular exercise over 30-60 minutes and complete 1-2 sets of 8 to 10 resistance/strength training exercises, 8 to 12 repetitions of each exercise, 3 days per week for 12 weeks. Patients also participate in weekly phone calls with an exercise physiologist to ensure adherence to the program and to provide support.
  Interventions: Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo resistance training program and cardiovascular exercise
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Participate in phone calls with exercise physiologist

SUMMARY:
This pilot trial studies how well a resistance training program and cardiovascular exercise work in increasing muscle mass in adolescent and young adult stem cell transplant survivors. Resistance training and cardiovascular exercise may increase physical activity, muscular strength and improve lean body mass which is beneficial to improving the overall health of stem cell transplant survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of a 12-week resistance training (RT) intervention in adolescent and young adult (AYA) hematopoietic cell transplant (HCT) survivors starting +100 days post-HCT.

SECONDARY OBJECTIVES:

I. Examine the change from baseline of a RT intervention on muscle strength and body composition at day +200 and day +365.

II. Determine the effectiveness of RT exercise on improving the cardio-metabolic risk factor profile at day +200 and day +365.

III. Determine the effectiveness of RT exercise on improving quality of life (QOL) measures.

IV. Compare day +80 and day +365 assessments to subjects in a historical control population.

OUTLINE:

Patients undergo moderately intense aerobic/cardiovascular exercise over 30-60 minutes and complete 1-2 sets of 8 to 10 resistance/strength training exercises, 8 to 12 repetitions of each exercise, 3 days per week for 12 weeks. Patients also participate in weekly phone calls with an exercise physiologist to ensure adherence to the program and to provide support.

After completion of study intervention, patients are followed up within 2 weeks, then at 365 days post HCT.

ELIGIBILITY:
Inclusion Criteria:

* > 80 days but less than <120 days post-autologous or allogeneic HCT for a malignancy.
* Platelet transfusion independent.
* Fully mobile on an independent basis.
* For patients who have been on steroid therapy for graft versus (vs) host disease, doses of prednisone must be =< 1.0 mg/kg/day and they must be on a tapering schedule.
* English speaking.

Exclusion Criteria:

* Individuals who are determined by the investigators or primary treating physician to not be physically able to participate in an independent exercise intervention such as hospitalized, wheel chair bound, unable to ambulate independently, on oxygen.
* Women who are pregnant will be excluded.

Ages: 13 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Enrollment rate | 200 Days
  Percentage of eligible, approached patients enrolling in program
Completion rate | At day +200 post hematopoietic cell transplant (HCT)
  Percentage of enrolled participants completing the full intervention
Adherence rate | At day +200 post hematopoietic cell transplant (HCT)
  Percentage of participants completing weekly follow-up phone calls

SECONDARY OUTCOMES:
Change in physical activity | Baseline to day +365 post HCT
  Measured using Actigraph activity monitor
Change in physical activity | Baseline to day +365 post HCT
  International Physical Activity Questionnaire (IPAQ)
Change in anthropometrics (BMI) | Baseline to day +365 post HCT
  Measured by BMI; weight and height will be combined to report BMI in kg/m^2
Change in cardiometabolic profile (Fasting Glucose, Insulin and Lipid Profile) | Baseline to day +365 post HCT
  Testing will be performed on patient blood samples. Changes will be calculated as score (approximately day +200) - score (approximately day+100). All variables will be described based on their distributions (means, standard deviations if normally distributed, medians and IQRs otherwise). A t-test will be used to compare means between baseline and follow-up time periods.
Heart rate | Baseline to day +365 post HCT
Change in body composition | Baseline to day +365 post HCT
  Measured using dual-energy x-ray absorptiometry (DXA). Changes will be calculated as score (approximately day +200) - score (approximately day+100). All variables will be described based on their distributions (means, standard deviations if normally distributed, medians and IQRs otherwise). A t-test will be used to compare means between baseline and follow-up time periods.
Change in muscular strength | Baseline to day +365 post HCT
  Strength testing will include hand grip strength, one repetition maximum chest press, one repetition maximum leg press and the 6 minute walk test. Changes will be calculated as score (approximately day +200) - score (approximately day +100). All variables will be described based on their distributions (means, standard deviations if normally distributed, medians and IQRs otherwise). A t-test will be used to compare means between baseline and follow-up time periods.
Blood pressure | Baseline to day +365 post HCT
Change in quality of life (QOL) | Baseline to day +365 post HCT
  Measured by the Patient-Reported Outcomes Measurement Information System
Incidence of adverse events | Up to day +200 post HCT

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Ketterl, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No